CLINICAL TRIAL: NCT02323594
Title: A Bioequivalence Study of the 90-mg Daclatasvir Tablet Relative to the 3 × 30-mg Daclatasvir Phase 3 Tablets, and Relative Bioavailability Studies of Chewable Pediatric Tablets of Daclatasvir and Asunaprevir in Healthy Adult Subjects
Brief Title: A Bioequivalence Study of Daclatasvir Tablets and Bioavailability Studies of Daclatasvir and Asunaprevir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AI447-111
Record Dates: First submitted 2014-12-09; First posted 2014-12-23 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; asunaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1: Daclatasvir (Experimental): Single oral dose of Daclatasvir (DCV) tablet and single oral dose of DCV pediatric chewable tablet
  Interventions: Drug: Daclatasvir
- Group 2: Daclatasvir (Experimental): Single oral dose of Daclatasvir (DCV) pediatric chewable tablet and single oral dose of DCV pediatric chewable tablet
  Interventions: Drug: Daclatasvir
- Group 3: Asunaprevir (Experimental): Single oral dose of Asunaprevir (ASV) tablet, single oral dose of ASV pediatric chewable tablet and single oral dose of ASV pediatric chewable tablets
  Interventions: Drug: Asunaprevir
- Group 4: Daclatasvir (Experimental): Single oral dose of Daclatasvir (DCV) tablet and single oral dose of DCV tablets
  Interventions: Drug: Daclatasvir

INTERVENTIONS:
Drug: Daclatasvir — Treatment A= single oral dose of Daclatasvir (DCV) tablet and Treatment B= single oral dose of DCV pediatric chewable tablet
  Arms: Group 1: Daclatasvir
Drug: Daclatasvir — Treatment C= single oral dose of Daclatasvir (DCV) pediatric chewable tablet and Treatment D= single oral dose of DCV pediatric chewable tablet
  Arms: Group 2: Daclatasvir
Drug: Asunaprevir — Treatment E= single oral dose of Asunaprevir (ASV) tablet and Treatment F= single oral dose of ASV pediatric chewable tablet and Treatment G= single oral dose of of ASV pediatric chewable tablet
  Arms: Group 3: Asunaprevir
Drug: Daclatasvir — Treatment H= single oral dose of Daclatasvir (DCV) tablet and Treatment I= single oral dose of DCV tablets
  Arms: Group 4: Daclatasvir

SUMMARY:
Grps 1, 2, 3 "This study will be testing the performance of ASV and DCV pediatric chewable tablets.

Grp #4 The purpose of this group is to support the marketing authorization of a DCV 90-mg tablet

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent must be obtained from the subjects in accordance with requirements of the study center's Institutional review Board (IRB)/ Institutional Ethics Committee (IEC)
2. Target Population: Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
3. Age and Reproductive Status : Males and females, ages 18 to 49 years, inclusive. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 24 hours prior to the start of study drug and must be using an acceptable method of contraception for 4 weeks prior to study drug administration. Women must not be breastfeeding.

Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for duration of treatment with study drug females must still undergo pregnancy testing as described in this section.

Exclusion Criteria:

1. Medical History and Concurrent Diseases : Any significant acute or chronic medical illness. Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug. Any major surgery within 4 weeks of study drug administration. Any gastrointestinal surgery that could impact upon the absorption of study drug (appendectomies with no complications are allowed at the investigator's discretion). Inability to tolerate oral medication, smokers or recent durg or alcohol abuse and Any other sound medical, psychiatric, and/or social reason as determined by the investigator.
2. Physical and Laboratory Test Findings: Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG, or clinical laboratory determinations beyond what is consistent with the target population, positive urine screen for drugs, positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or HIV-1, -2 antibodies.
3. Allergies and Adverse Drug Reaction : History of allergy to DCV, ASV, Hepatitis C virus (HCV) NS3 protease inhibitors, HCV NS5A replication cofactors, or related compounds.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration [Cmax] | Before dosing through 96 hours
Area under the concentration-time curve [AUC] from time zero extrapolated to infinite time [AUC(INF)] | Before dosing through 96 hours
AUC from time zero to the time of last quantifiable concentration [AUC(0-T)] | Before dosing through 96 hours
Time of maximum observed plasma concentration [Tmax] | Before dosing through 96 hours
Terminal plasma half life [T-HALF]) | Before dosing through 96 hours

SECONDARY OUTCOMES:
Adverse Event reports | 30 days after last dose
  Safety assessments based on review of adverse events, vital sign measurements, electrocardiograms, physical examinations, and clinical laboratory tests.
Vital sign measurements | 30 days after last dose
ECGs | 30 days after last dose
Physical examinations | 30 days after last dose
Clinical laboratory tests | 30 days after last dose
The incidence of reported AEs will be tabulated and reviewed for potential significance and clinical importance. | 30 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca N Wood-Horrall, MD, Principal Investigator — PPD Development, LP